CLINICAL TRIAL: NCT06324942
Title: Analgesic Efficacy of Surgeon-administered Transversus Abdominis Plane Blocks for Caesarean Section.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Stephen Wood, Dr Stephen Wood, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB24-0349
Record Dates: First submitted 2024-03-07; First posted 2024-03-22 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Cesarean Section Complications; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgeon-administered Transversus Abdominis Plane Block (TAP block) (Experimental): After uterine closure, the anterior abdominal wall on the contralateral side to the surgeon is elevated and retracted laterally by an assistant. The bowel and uterus is retracted using the surgeon's non-dominant hand, with or without a sponge. Under direct visualization, a blunted spinal needle is inserted lateral to the rectus muscle to avoid injury to inferior epigastric blood vessels. The needle is then gently advanced through the transversus abdominis fascia into the TAP plane, identified at loss of resistance, or 'a pop'. After aspiration to confirm no accidental placement of the needle intravascularly, local anaesthetic is infiltrated into the transverse abdominis plane through the parietal peritoneum by the surgeon at a prespecified dose of 0.25% bupivicaine 0.25 mL/kg (approximately 20cc). This is repeated on the contralateral side, after which closure of the fascia, subcutaneous tissue, and skin were performed.
  Interventions: Other: Surgeon-administered Transversus Abdominis Plane Block 0.25% bupivicaine 0.25 mL/kg
- No TAP block (No Intervention): A sham procedure will not be performed but the patient will be unaware of whether or not an injection was done.

INTERVENTIONS:
Other: Surgeon-administered Transversus Abdominis Plane Block 0.25% bupivicaine 0.25 mL/kg — Surgeon-administered Transversus Abdominis Plane Block
  Other Names: TAP block
  Arms: Surgeon-administered Transversus Abdominis Plane Block (TAP block)

SUMMARY:
The purpose of this research study is to evaluate whether or not adding a Transversus Abdominis Plane Block (TAP block) improves pain control for patients having a cesarean section. A TAP block is a type of nerve block where at the end of the surgery an injection of a long acting local anesthetic is made into the abdominal wall. In studies in patient's having other abdominal surgeries this has reduced the amount of narcotics patients need for pain control. This may also led to patients being more active after surgery and maybe spending less time in hospital.

DETAILED DESCRIPTION:
Randomized clinical trial of Transversus Abdominis Plane Block (TAP block) at Cesarean Section.

ELIGIBILITY:
Inclusion Criteria:

* ASA status II to III
* All patients undergoing elective CS under regional anesthesia at any gestational age.

Exclusion Criteria:

* - Known drug allergy to local anesthetics
* Planned general anesthetic
* NSAID use contraindicated post partum
* Chronic pain disorder or chronic narcotic use/dependence
* Planned vertical abdominal incision
* Planned Cesarean Hysterectomy.
* Placenta Previa or suspected Placenta Accreta

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Post operative Pain | 12 hours post op
  VAS scale 0-no pain to 10-worst pain

SECONDARY OUTCOMES:
Time to first request for rescue analgesia in hours | 48 hours post op
  Time from completion of surgery to first request for rescue analgesia in hours
Post operative Opioid use | up to 48 hours post op.
  Total opioid consumption in the first 24h and 48h mark, postoperatively
Time from surgery to discharge from hospital | Up to discharge from hospital, usually 1-3 days
  Time from completion of surgery to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Wood, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT06324942/Prot_SAP_000.pdf